CLINICAL TRIAL: NCT02417623
Title: Efficacy of a Mobile Application for Weight Loss in Overweight and Obese Adults: A Randomized Controlled Trial
Brief Title: Smartphone Application for Weight Loss
Acronym: OBSBIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/07 IDIAP
Record Dates: First submitted 2015-03-26; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smartphone intervention group (Experimental): The experimental group will receive the standard diet intervention for weight loss plus free Smartphone app plus a wearable device.
  Interventions: Behavioral: Smartphone Application group
- Control group (No Intervention): Control group will receive a 12-month weight loss programmed that implements recommendations of a Clinical Practice Guideline

INTERVENTIONS:
Behavioral: Smartphone Application group — Intervention group will receive a 12-month weight loss programmed that implements recommendations of a Clinical Practice Guideline, complemented with a smartphone app
  Arms: Smartphone intervention group

SUMMARY:
AIM: To assess the efficacy of an intervention that includes the assistance of a weight loss smartphone application targeted to young people aged 18 to 40 years.

DESIGN: Randomisedclinical trial.

SETTING: Primary Health Care centres (PHCCs) in Catalonia.

PARTICIPANTS: Adults aged 18 to 40 years with criteria of obesity or overweight, consulting PHCCs for any reason and who provide written informed consent to participate in the trial.

INTERVENTION GROUP will receive a 12-month weight loss programme that implements recommendations of a Clinical Practice Guideline, complemented with a smartphone app designed specifically for this programme.

CONTROL GROUP will receive the usual care. The outcome measure will be weight loss at 12 months.

EXPECTED RESULTS: The investigators expect a higher weight loss in the intervention group than in control group.

DETAILED DESCRIPTION:
DESIGN: Randomised clinical trial.

SETTING: Primary Health Care centres (PHCCs) in Catalonia, Spain.

PARTICIPANTS: Adults aged 18 to 40 years with criteria of obesity or overweight, consulting PHCCs for any reason and who provide written informed consent to participate in the trial.

INTERVENTION GROUP will receive a 12-month weight loss programme that implements recommendations of a Clinical Practice Guideline, complemented with a smartphone app designed specifically for this programme.

CONTROL GROUP will receive the usual care. The outcome measure will be weight loss at 12 months.

EXPECTED RESULTS: The investigators expect a higher weight loss in the intervention group than in control group.

ELIGIBILITY:
Inclusion Criteria:

* Young adults aged 18 to 40 years with overweight or obesity
* availability of the patient's clinical history in the primary care centre
* access to a smartphone device that meets the app requirements
* access to an Internet data connection

Exclusion Criteria:

* Morbid obesity with BMI> 40
* Secondary Obesity (eg endocrine pathology)
* eating disorders (the patient or any member of the family);
* Presence of any significant comorbidity that a specific treatment (type 1 diabetes mellitus, severe mental illness);
* pregnant or desire pregnancy in the next 12 months;
* To participate in a weight loss program or taking any medication for weight loss in the moment of the recruitment
* Take any medication that may influence body weight;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Body weight (Kg) | 12 months
  Change in body weight at 12 months in the experimental group, compared with the control group. At each study visit, anthropometrics will be recorded by a primary care nurse or doctor. Body weight will be measured with the participant dressed in light clothing with shoes off on a calibrated balance.
Body mass index (Kg/m2) | 12 months
  change in body mass index at 12 months in the experimental group, compared with the control group.. At each study visit, anthropometrics will be recorded by a primary care nurse or doctor. Body weight will be measured with the participant dressed in light clothing with shoes off on a calibrated balance.

SECONDARY OUTCOMES:
Physical activity measured with two brief validated questionnaires | 12 months
  To increase physical activity at 12 months. Physical activity will be measured with two brief validated questionnaires, administered in the participant's preferred language (Catalan or Spanish).
glucemic levels | 12 months
  To improve the glucose levels
cholesterol profile (LDL-cholesterol, HDL-Cholesterol, Cholesterol total) | 12 months
  To improve the profile of cholesterol.
blood pressure | 12 months
  To improve the blood pressure
GPT levels | 12 months
  To monitorize GPT levels

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Health Care La Granja- Torreforta, Tarragona, Spain

REFERENCES:
- [Derived] Granado-Font E, Flores-Mateo G, Sorli-Aguilar M, Montana-Carreras X, Ferre-Grau C, Barrera-Uriarte ML, Oriol-Colominas E, Rey-Renones C, Caules I, Satue-Gracia EM; OBSBIT Study Group. Effectiveness of a Smartphone application and wearable device for weight loss in overweight or obese primary care patients: protocol for a randomised controlled trial. BMC Public Health. 2015 Jun 4;15:531. doi: 10.1186/s12889-015-1845-8. PMID 26041131